CLINICAL TRIAL: NCT04138589
Title: Real World Data of the Effect of Lumacaftor/Ivacaftor Therapy in Children With Cystic Fibrosis Homozygote for F508del on Small Airway Function
Brief Title: Effect of Lumacaftor/Ivacaftor in Children With Cystic Fibrosis Homozygote for F508del on Small Airway Function
Acronym: ROOTS
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry); Marien Hospital Wesel (Other)
Responsible Party: Principal Investigator, A.M. Zwitserloot, MD, University Medical Center Groningen
Other Study IDs: 201900032
Record Dates: First submitted 2019-09-18; First posted 2019-10-24 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis in Children
Keywords: lumacaftor/ ivacaftor; tezacaftor/ ivacaftor; Multiple breath washout; Lung clearance index; PRAGMA CF score

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CF patients aged 6-18 years homozygeous for delta F508: CF patients aged 6-18 years homozygeous for delta F508 starting with lumacaftor/ ivacaftor or tezacaftor/ ivacaftor

SUMMARY:
To obtain prospective real world data of the effect of lumacaftor/ivacaftor or tezacaftor/ ivacaftor on small airway disease in children aged 6-18 years with cystic fibrosis (CF) homozygous for F508del. The effect of the medication on small airway disease is evaluated by measurement of multiple breath washout (MBW) with its outcome parameter lung clearance index (LCI) and the Perth-Rotterdam Annotated Grid Morphometric Analysis for CF (PRAGMA-CF) cpmputed tomography (CT) score. In addition the relation between changes in LCI and PRAGMA-CF score is evaluated.

DETAILED DESCRIPTION:
Multi-center observational study. Duration 12 months after the start of lumacaftor/ ivacaftor or tezacaftor/ ivacaftor .

To collect these data and to assist in clinical decisions regarding initiation and continuation of lumacaftor/ivacaftor or tezacaftor/ ivacaftor, the investigators of the CF center (Beatrix Children's Hospital, University Medical Center Groningen (UMCG), the Netherlands) developed an extensive protocol of testing before children aged 6-18 years start therapy and during the first year after start.

The protocol includes the following tests: growth parameters, sweat test, lung function testing (spirometry, MBW, body plethysmography), blood test panel (AST, ALT, alkalic phosphatase (AF), total and direct bilirubin, LDH), fecal elastase, high resolution (HR)CT and CF quality of life questionnaires. These tests are repeated at regular intervals.

Multi-center observational study. Duration 12 months after the start of lumacaftor/ ivacaftor or tezacaftor/ ivacaftor .

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-18 years
* CF, Homozygote F508del confirmed by DNA analysis
* Considered for start of lumacaftor/ ivacaftor or tezacaftor/ivacaftor

Exclusion Criteria:

* - Unable to perform acceptable, repeatable lung function tests

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients are included from the Beatrix Children's Hospital, UMCG, the Netherlands and the Marien Hospital Wesel, Germany
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Change in lung clearance index | 12 months
  Change between t=0 and t=12

SECONDARY OUTCOMES:
Change in PRAGMA-CF score | 12 months
  Change between t=0 and t=12

OTHER OUTCOMES:
percent predicted forced expiratory volume in 1 second | 12 months
  t= 0 and t-=12
percent predicted forced vital capacity measured by spirometry | 12 months
  Change between t=0 and t=12
Residual volume measured by blodypethysmography | 12 months
  Change between t=0 and t=12
Residual volume/ total lung capacity measured by blodypethysmography | 12 months
  Change between t=0 and t=12
Mid upper arm circumference in SDS | 12 months
  Change between t=0 and t=12
Weight SDS | 12 months
  Change between t=0 and t=12
Sweat chloride level | 12 months
  Change between t=0 and t=12
CF questionnaire revised respiratory domain | 12 months
  Change between t=0 and t=12, scale 0-100

CONTACTS AND LOCATIONS:
Locations (2):
- Children's Hospital Marien Hospital Wesel, Düsseldorf, Germany
- Beatrix Children's Hospital, University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD